CLINICAL TRIAL: NCT00967135
Title: Efficacy of Perioperative Pregabalin in Reducing the Incidence of Chronic Neuropathic Pain and Postthoracotomy Syndrome.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PC 2010-001
Record Dates: First submitted 2009-08-26; First posted 2009-08-27 (Estimated); Last update posted 2012-04-12 (Estimated); Status verified 2012-04

CONDITIONS: Neuropathic Pain
Keywords: Thoracotomy; Neuropathic pain
MeSH Terms: conditions — Neuralgia | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pregabalin (Experimental): Study subjects will be randomized to receive on the morning of surgery, at least 30 minutes before induction, a 150 mg oral dose of pregabalin. Patients will then receive a 150 mg oral dose of pregabalin on the evening of the surgery. Subsequently, patients will receive a 150 mg oral dose of pregabalin twice daily on the following four postoperative days.
  Interventions: Drug: Pregabalin
- Placebo (Placebo Comparator): Study subjects will be randomized to receive a matching placebo on the morning of surgery, at least 30 minutes before induction. Patients will then receive a placebo on the evening of the surgery. Subsequently, patients will receive a placebo twice daily on the following four postoperative days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pregabalin — 150 mg oral dose of pregabalin twice daily for 5 consecutive days.
  Other Names: Lyrica
  Arms: Pregabalin
Drug: Placebo — Matching oral placebo twice daily for 5 consecutive days.
  Arms: Placebo

SUMMARY:
This study is designed to assess:

1. The impact of taking perioperative pregabalin on the incidence of chronic neuropathic pain and postthoracotomy syndrome at 3 months in patients who have undergone a thoracotomy with a thoracic epidural as the basic analgesic modality.
2. The impact of taking perioperative pregabalin on the relief of acute pain, and on the use of additional analgesics, such as opioids, for the relief of such pain in patients who have undergone thoracic surgery with a thoracic epidural as the basic analgesia.
3. The impact of taking perioperative pregabalin on the quality of life and level of functioning of patients who underwent thoracic surgery 3 months earlier.
4. The safety profile of pregabalin in this patient population.

Hypothesis: The basic hypothesis in this study is that a dose of pregabalin administered preemptively 1 hour before a thoracotomy, then repeatedly during the postoperative period, when neuronal hyperexcitability is at a maximum (i.e., 4 days), will lead to a 33.3% decrease in the prevalence of chronic pain 3 months after surgery.

DETAILED DESCRIPTION:
Postthoracotomy pain syndrome is a rather frequent phenomenon. Its incidence, as reported in the literature, varies but is around 52% at 1 to 2 years after surgery. This syndrome is defined as a persistent and/or recurrent pain or burning sensation along the thoracotomy scar at least 2 months after surgery. The pain is very significant, given that 3 to 5% of patients report it as being severe, and approximately 50% of patients report limitations in their activities of daily living secondary to this pain and consider their pain as their worst medical problem. A neuropathic component makes a certain contribution to this pain. Patients with this neuropathic component report more-severe pain and take more analgesics. Little is known about the origin of this pain, but it seems that the intensity of acute postoperative pain is the best predictor of it. Pregabalin could be a possible approach to reducing the prevalence of chronic postthoracotomy pain. Its efficacy has been demonstrated in several diabetic, postherpetic, incisional and inflammatory neuropathic pain models.

Methods:

One hundred and twenty patients will be divided in two equal groups (to receive pregabalin or placebo).

Prior to the induction of general anesthesia, a thoracic epidural will be placed and started immediately prior to surgery. The anesthetic technique and monitoring will be standardized.

During the immediate postoperative period, the intensity of pain will be assessed using a VNPS (0-10). Pain will be assessed upon the patient's arrival in and discharge from the recovery room and daily thereafter, for a total duration of four postoperative days or until discharge from hospital if this occurs before the 4th postoperative day.

Three months after their surgery, the patients will be contacted by telephone and administered a standardized questionnaire for evaluating:

* The presence and intensity (based on a VNPS) of pain at the surgical and/or drainage tube sites.
* The type of pain, with specific attention to identifying the presence of neuropathic pain.
* The patients' assessment of their quality of life, and the impact, if any, of the pain on their level of functioning in their daily lives in relation to their preoperative quality of life and functioning.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 80 years.
* Patients who are to undergo an elective thoracotomy in the lateral decubitus position.
* Patients who are ASA I to III inclusive.

Exclusion Criteria:

* A contraindication to pregabalin.
* A contraindication to the epidural technique.
* The current use of drugs belonging to the class of opioids, NMDA receptor blockers, membrane stabilizing agents (lidocaine mesylates, flecainide) or topical coanalgesics (capsaicin cream, lidocaine patch).
* Previous use of pregabalin or gabapentin.
* Preexisting pain at the site where the surgical incision will be made.
* Presence of a coexisting chronic pain syndrome.
* A creatinine clearance of less than 60 mL/min.
* A previous ipsilateral thoracotomy.
* A recent history of alcohol and/or drug abuse.
* A known allergy to local anesthetics or hydromorphone.
* The inability to understand a verbal numerical pain scale (VNPS) despite previous instruction.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2010-06; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Development of neuropathic pain and intensity of pain assessed using the Leeds Assessment of Neuropathic Symptoms and Signs (LANSS) scale and Brief Pain Inventory questionnaire (BPI). | At 3 months

SECONDARY OUTCOMES:
Intensity of postoperative pain using a Visual Numeric Pain Scale (VNPS). | Day 1 to Day 4

CONTACTS AND LOCATIONS:
Overall Officials: François Girard, MD, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre Hospitalier de l'Université de Montréal (Hôpital Notre-Dame), Montreal, Quebec, Canada